CLINICAL TRIAL: NCT02312674
Title: Prevention of Malnutrition Through Oral Nutritional Supplements in Cancer Patients Receiving Palliative Therapy
Brief Title: Prevention of Cancer-associated Malnutrition Through Oral Nutritional Supplements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Hohenheim (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZEM_Minigrad_TN
Record Dates: First submitted 2014-11-07; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-11

CONDITIONS: Cancer
Keywords: pancreatic carcinoma; hepatocellular carcinoma; palliative therapy; oral nutritional supplements; quality of life; nutritional status
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Carcinoma, Hepatocellular | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patient group which takes daily an adjusted amount of oral nutritional supplements through an intervention period of three months
  Interventions: Dietary Supplement: Oral nutritional supplement
- Control (No Intervention): Patients group which takes no oral nutritional supplements

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement — Beginning with the start of palliative therapy, depending on the nutritional status, one, two, or three cans per day are ingested during a period of three months.
  Other Names: Fortimel Compact/Fortimel Compact Fibre, Nutricia
  Arms: Intervention

SUMMARY:
The aim of the randomized controlled study is to determine effects of an adjusted amount of oral nutritional supplements on the quality of life, the nutritional status, side effects, and response to therapy, in patients with pancreatic and hepatocellular carcinoma receiving palliative therapy.

DETAILED DESCRIPTION:
Cancer is often associated with malnutrition and weight loss. The occurence of malnutrition during the course of the disease depends on the type, extent, and therapy of the tumor. Pancreatic cancer patients and patients with hepatocellular carcinoma are particularly at risk of developing a pronounced weight loss. Cancer-related malnutrition has negative impact on the response to therapy, survival, quality of life, and the infection rate of patients, resulting in prolonged hospital stays and higher costs for health care. Maintaining or optimizing the quality of life in patients receiving palliative therapy has priority. Since a poor nutritional status affects the quality of life, patients might benefit from the use of an adjusted amount of oral nutritional supplements.

To determine the effects of oral nutritional supplements, a controlled randomized study will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* assured diagnosis of pancreatic cancer/hepatocellular carcinoma, not treatable with curative intent
* palliative systemic therapy of pancreatic cancer respectively palliative therapy of hepatocellular carcinoma with Sorafenib or TACE (transarterial chemoembolization)
* written informed consent prior to inclusion

Exclusion Criteria:

* prefinal phase with an estimated life expectancy of less than three months
* nutritional support through tube feeding or a central venous catheter
* serious malassimilation (assessed by anamnesis)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≥ 2
* hepatic encephalopathy ≥ degree 2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life | Every four weeks for a period of three months and after six months
  Health-related quality of life is assessed by using the standardized questionnaire "Short Form-36 Health Survey" (SF36).
Change in disease-related quality of life | Every four weeks for a period of three months and after six months
  Disease-related quality of life is assessed by using the standardized questionnaire "Functional Assessment of Cancer Therapy - Hepatobiliary questionaire" (FACT-Hep).

SECONDARY OUTCOMES:
Body mass index (BMI) | Every four weeks for a period of three months and after six months
  To calculate the BMI, weight and height are measured.
Body composition | Every four weeks for a period of three months and after six months
  To measure the body composition, a bioelectrical impedance analysis (BIA) is carried out. The phase angle and the extracellular cell mass/body cell mass ratio (ECM/BCM ratio) is evaluated.
Grip strength [lb] | Every four weeks for a period of three months and after six months
  To measure the grip strength, a hydraulic force measuring device is used.
Score (points) of nutritional risk screening | Every four weeks for a period of three months and after six months
  Patients are screened with the Nutritional Risk Screening 2002 (NRS 2002)
Laboratory parameters | Every four weeks for a period of three months and after six months
  Albumin, C-reactive protein (CRP), Ferritin are measured to assess the nutritional and protein status as well as the disease activity

OTHER OUTCOMES:
Average daily energy intake [kcal] | Every four weeks for a period of three months and after six months
  To assess the average daily energy intake patients keep a food diary over two days between the trial dates
Side effect profile | Every four weeks for a period of three months and after six months
  The occurrence and extent of tumor-associated and nutritional therapy-associated side effects are determined using Common Terminology Criteria for Adverse Events (CTCAE)
Dose density | After three months
  The dose density is determined by the intended and actual administered respectively ingested dose of medication. The dose density is taken from the chemotherapy protocols or determined based on taking notes.
Tumor response | After three months
  In patients with pancreatic cancer tumor staging is performed based on the Response Evaluation Criteria in Solid Tumors (RECIST criteria), in patients with hepatocellular carcinoma tumor staging is performed based on the modified RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, MD, Prof., Principal Investigator — Department of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany; Michael Bitzer, MD; Prof., Study Director — Department of Hepatology, Gastroenterology, Infectious Diseases, University Hospital Tübingen